CLINICAL TRIAL: NCT00153166
Title: The Contribution of Inflammation and Insulin Resistance to Intermittent Claudication
Brief Title: ARREST PAD (Peripheral Arterial Disease)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mark Alan Creager, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003P-001501; R01HL075771 (NIH); NCT00225940 (obsolete NCT alias)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Arterial Occlusive Disease; Intermittent Claudication; Insulin Resistance
Keywords: peripheral arterial disease; intermittent claudication
MeSH Terms: conditions — Arterial Occlusive Diseases; Intermittent Claudication; Insulin Resistance; Peripheral Arterial Disease | interventions — Atorvastatin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patients with PAD (Including diabetics) (Experimental): Randomized to either atorvastatin and pioglitazone, atorvastatin/placebo, pioglitazone/placebo, or placebo/placebo.
  Interventions: Drug: atorvastatin and pioglitazone; Drug: atorvastatin/placebo; Drug: pioglitazone/placebo; Drug: placebo/placebo
- PAD (Excluding Diabetics) (Active Comparator): Randomized to either atorvastatin and pioglitazone, atorvastatin/placebo, pioglitazone/placebo, or placebo/placebo.
  Interventions: Drug: atorvastatin and pioglitazone; Drug: atorvastatin/placebo; Drug: pioglitazone/placebo; Drug: placebo/placebo
- Healthy Controls (Active Comparator): Randomized to either atorvastatin and pioglitazone, atorvastatin/placebo, pioglitazone/placebo, or placebo/placebo.
  Interventions: Drug: atorvastatin and pioglitazone; Drug: atorvastatin/placebo; Drug: pioglitazone/placebo; Drug: placebo/placebo

INTERVENTIONS:
Drug: atorvastatin and pioglitazone — atorvastatin 80 mg orally once daily (to reduce inflammation) and pioglitazone 30 mg orally once daily (to improve insulin sensitivity)
  Other Names: atorvastatin: lipitor; pioglitazone: actos
Drug: atorvastatin/placebo — atorvastatin 80 mg orally once daily and matching placebo orally twice daily
  Other Names: atorvastatin: lipitor
Drug: pioglitazone/placebo — pioglitazone 30 mg orally once daily and matching placebo orally once daily
  Other Names: pioglitazone: actos
Drug: placebo/placebo — placebo orally three times daily

SUMMARY:
This trial will test the hypothesis that inflammation and insulin resistance contribute to reduced walking distance in subjects with intermittent claudication by impairing vascular reactivity and skeletal muscle metabolic function.

DETAILED DESCRIPTION:
People with peripheral arterial disease (PAD), an important clinical manifestation of atherosclerosis, often suffer symptoms of intermittent claudication that impair their walking ability and adversely affect their quality of life. People with PAD are also at increased risk for adverse cardiovascular events, including myocardial infarction, stroke and death. Unfortunately, medical therapies directed to the functional and limb-threatening manifestations are limited. Little attention has been paid to the biologic processes that cause PAD, and to atherogenic mechanisms that may preferentially affect the peripheral circulation.

Vascular inflammation and insulin resistance are two important and interdependent conditions that are associated with atherosclerosis. Subjects in this trial (160 adults with stable intermittent claudication who are not taking insulin or insulin-sensitizing medications, such as thiazolidinediones) will be randomized in a placebo-controlled, parallel design manner, to atorvastatin 80 mg orally daily (to reduce inflammation) and pioglitazone 45 mg orally once daily (to improve insulin sensitivity). Forty healthy adult subjects, age and gender-matched to a subset of the study group, will be enrolled to serve as a control population. Primary and secondary study endpoints include: treadmill walking time, endothelium-dependent vasodilation, and insulin-mediated skeletal muscle glucose uptake.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic intermittent claudication for >= 6 months
* resting ankle/brachial index (ABI) <=0.90
* maximal treadmill walking time between 1-20 minutes
* >= 20% decrease in ABI post treadmill exercise
* 4 week statin wash-out prior to initial study testing (if applicable)

Exclusion Criteria:

* myocardial infarction or coronary artery bypass surgery within past 6 months
* lower extremity revascularization (surgical or percutaneous) within past 6 months
* transient ischemic attack or ischemic stroke within past 6 months
* pregnancy
* uncontrolled hypertension (systolic pressure > 180mmHg and/or diastolic pressure > 100mmHg
* serum creatinine >2.5
* hepatic transaminases (AST, ALT) > 3x upper limit of normal (ULN)
* creatine kinase > 5x ULN
* known hypersensitivity to HMG-CoA reductase inhibitors
* insulin dependent Type 2 diabetes
* current treatment with thiazolidinedione

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-01; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Creager, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Pande RL, Brown J, Buck S, Redline W, Doyle J, Plutzky J, Creager MA. Association of monocyte tumor necrosis factor alpha expression and serum inflammatory biomarkers with walking impairment in peripheral artery disease. J Vasc Surg. 2015 Jan;61(1):155-61. doi: 10.1016/j.jvs.2014.06.116. Epub 2014 Aug 2. PMID 25095746

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Healthy individuals, non-smokers, normal CV examination. Randomized to atorvastatin/pioglitazone, atorvastatin/placebo, placebo/pioglitazone, or placebo/placebo.
- Patients With PAD: Patients with PAD and stable intermittent claudication with a resting ABI of 0.90 or less. Randomized to atorvastatin/pioglitazone, atorvastatin/placebo, placebo/pioglitazone, or placebo/placebo.
- PAD (Excluding Patients With Diabetes): Patients with PAD and stable intermittent claudication with a resting ABI of 0.90 or less. Excluding those patients with diabetes. Randomized to atorvastatin/pioglitazone, atorvastatin/placebo, placebo/pioglitazone, or placebo/placebo.
Period: Overall Study
Arm/Group | Healthy Controls | Patients With PAD | PAD (Excluding Patients With Diabetes)
Started | 11 | 37 | 28
Received Atorvastatin and Pioglitazone | 3 | 9 | 7
Received Atorvastatin and Placebo | 2 | 9 | 7
Received Placebo and Pioglitazone | 3 | 10 | 7
Received Placebo and Placebo | 3 | 9 | 7
Completed | 11 | 37 | 28
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were collected according to the clinical diagnosis of the patients and not according to randomization. Participants are grouped at Baseline regardless of randomization because we are measuring baseline characteristics that do not depend on which intervention they received.
Groups:
- Healthy Controls: Healthy individuals, non-smokers, normal CV examination.
- Patients With PAD: Patients with PAD and stable intermittent claudication with a resting ABI of 0.90 or less.
- PAD Without Diabetes: Patients with PAD and stable intermittent claudication with a resting ABI of 0.90 or less. These patients do not have diabetes.
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Patients With PAD | PAD Without Diabetes | Total
Number analyzed (Participants) | 11 | 37 | 28 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 6 | 15
  >=65 years | 8 | 31 | 22 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (6) | 66 (8.7) | 64.6 (8.8) | 64.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 15
  Male | 5 | 31 | 25 | 61
Region of Enrollment [Number; unit: participants]
  United States | 11 | 37 | 28 | 76

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Skeletal Muscle Glucose Uptake
Description: Net calf skeletal muscle glucose uptake determined by Patlak modeling.
Time Frame: 60 minutes
Population: Baseline Characteristics were collected according to the clinical diagnosis of the patients and not according to randomization. Participants were grouped at Baseline and are presented here irrespective of randomization because the primary intention was to compare the different types of patients regardless of interventions received.
Measure: Mean (Standard Deviation); unit: umol/kg/min
Groups:
- PAD (Excluding Diabetes): Patients with PAD and stable intermittent claudication with a resting ABI of 0.90 or less. These patients do not have diabetes.
Arm/Group | Healthy Controls | Patients With PAD | PAD (Excluding Diabetes)
Number analyzed (Participants) | 11 | 37 | 28
umol/kg/min | 62.9 (21) | 48.6 (15) | 49.5 (3.1)

2. Secondary Outcome: 'M' = Whole Body Insulin Sensitivity
Description: A hyperinsulinemic-euglycemic clamp was performed prior to and during FDG-PET imaging to measure insulin sensitivity and to standardize metabolic conditions. Subjects were required to fast for 8 hours prior to the study. Patients were given a primed insulin infusion of 2 mU/kg/min. Serum glucose measurements were made at five-minute intervals from an arterialized venous sample achieved by placing the hand in a warming box at 50°C. Blood glucose levels are checked every 5 minutes and 20% dextrose infusion is adjusted to maintain a serum glucose level of approximately 80 mg/dL. Subjects were considered to have achieved steady state when the dextrose infusion rate required to maintain a serum glucose level of 80 mg/dL varied by no greater than 5%. To compute the steady-state glucose disposal rate, we averaged the glucose infusion rates over the last 20 minutes of the clamp and applied a "space correction" to account for small changes in serum glucose levels over that time period.
Time Frame: every 5 minutes for 20 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Arm/Group | Healthy Controls | Patients With PAD | PAD (Excluding Diabetes)
Number analyzed (Participants) | 11 | 37 | 28
mg/kg/min | 5.0 [3.7 to 6.6] | 3.4 [2.7 to 4.8] | 3.4 [2.8 to 4.9]

ADVERSE EVENTS:
Groups:
- Received Atorvastatin/Pioglitazone; Received Atorvastatin/Placebo; Received Placebo/Pioglitazone; Received Placebo/Placebo: Including healthy subjects and subjects with PAD
Arm/Group | Received Atorvastatin/Pioglitazone | Received Atorvastatin/Placebo | Received Placebo/Pioglitazone | Received Placebo/Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No